CLINICAL TRIAL: NCT02345382
Title: An Open-label Phase I Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of BAY1143572 Given in a Once-daily or an Intermittent Dosing Schedule in Subjects With Advanced Acute Leukemia
Brief Title: Phase I Dose Escalation of BAY1143572 in Subjects With Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16520; 2014-000410-57 (EudraCT Number)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Leukemia
Keywords: Advanced acute leukemia
MeSH Terms: conditions — Leukemia | interventions — atuveciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 20 mg BAY1143572 (Experimental): Subjects received 20 milligram (mg) BAY1143572 tablet orally once daily from Cycle 1 Day 1 of each cycle.
  Interventions: Drug: Atuveciclib, BAY1143572
- 40 mg BAY1143572 (Experimental): Subjects received 40 mg BAY1143572 tablet orally once daily from Cycle 1 Day 1 of each cycle.
  Interventions: Drug: Atuveciclib, BAY1143572
- 80 mg BAY1143572 (Experimental): Subjects received BAY1143572 80 mg tablet orally once daily from Cycle 1 Day 1 of each cycle.
  Interventions: Drug: Atuveciclib, BAY1143572
- 120 mg BAY1143572 (Experimental): Subjects received BAY1143572 120 mg tablet orally once daily from Cycle 1 Day 1 of each cycle.
  Interventions: Drug: Atuveciclib, BAY1143572
- 160 mg BAY1143572 (Experimental): Subjects received BAY1143572 160 mg tablet orally once daily from Cycle 1 Day 1 of each cycle.
  Interventions: Drug: Atuveciclib, BAY1143572
- 200 mg BAY1143572 (Experimental): Subjects received BAY1143572 200 mg tablet orally once daily from Cycle 1 Day 1 of each cycle.
  Interventions: Drug: Atuveciclib, BAY1143572
- 240 mg BAY1143572 (Experimental): Subjects received BAY1143572 240 mg tablet orally once daily from Cycle 1 Day 1 of each cycle.
  Interventions: Drug: Atuveciclib, BAY1143572

INTERVENTIONS:
Drug: Atuveciclib, BAY1143572 — The starting dose was 20 mg BAY 1143572 once daily from Cycle 1 Day 1. Each cycle was defined as a period of 28 days. Dosing cycles continued until evidence of progression, unacceptable toxicity, consent withdrawal, or withdrawal from the study at the discretion of the investigator.

SUMMARY:
To determine the safety, tolerability, pharmacokinetics, maximum tolerated dose, and recommended Phase II dose of BAY1143572 in a once-daily or an intermittent dosing schedule in subjects with advanced acute leukemia

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged >/=18 years
* Subjects with a histologically or cytologically confirmed acute leukemia who are refractory to or have exhausted all available therapies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy of at least 12 weeks
* Adequate liver and renal functions as assessed by the following laboratory requirements to be conducted within 14 days before the first dose of study drug:

  * Total bilirubin </=1.5 times the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </=2.5 times ULN (</=5 times ULN for subjects with liver involvement of their cancer)
  * International normalized ratio (INR) </=1.5 times ULN
  * Estimated glomerular filtration rate (eGFR) >/=50 mL/min per 1.73 m2 according to the Modification of Diet in Renal Disease Study Group (MDRD) formula
* Negative serum or urine pregnancy test must be obtained within 7 days before the first dose of study drug in women of childbearing potential. Negative results must be available before study drug administration
* Women and men of reproductive potential must agree to use highly effective contraception when sexually active. This applies for the period between signing of the informed consent and 30 days after the last administration of study drug. Highly effective contraception includes a hormonal contraception with implants or combined oral contraceptives, certain intrauterine devices, bilateral tubal ligation, hysterectomy, or vasectomy of the partner. In addition, the use of condoms for subjects or their partners is required.

Exclusion Criteria:

* Known hypersensitivity to the study drug or excipients of the preparation or any agent given in association with this study
* History of cardiac disease including congestive heart failure New York Heart Association (NYHA) Class >/=III, unstable angina (anginal symptoms at rest) or new-onset angina (within the last 6 months) or myocardial infarction within the past 6 months or cardiac arrhythmias requiring anti-arrhythmic therapy except for beta-blockers and digoxin; evidence for uncontrolled coronary artery disease (e.g. major regional wall motion abnormalities on baseline echocardiography or a left ventricular ejection fraction (LVEF) <45%)
* Previous pulmonary embolism within 12 months before study entry
* Uncontrolled hypertension defined as systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg, despite optimal medical management and stable antihypertensive treatment for more than 7 days before the first dose of study drug
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C
* Known history of human immunodeficiency virus (HIV) infection
* Chronic or active hepatitis B or C, requiring antiviral therapy
* Serious, uncontrolled infection requiring systemic antibiotic, antifungal or antiviral therapy
* Uncontrolled meningeal leukemia
* Prior allogeneic hematopoietic stem cell transplant within </=4 months before first dose of study drug (Subjects must have completed immunosuppressive therapy before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of BAY1143572 in Advanced Acute Leukemia Subjects | After the first 28 days of treatment (cycle 1)
  The MTD was defined as the highest dose that could be given such that not more than 20% of subjects experience a dose limiting toxicity (DLT) during Cycle 1. The study was terminated prior to the determination of MTD and hence no data was presented.
Maximum Total Observed Drug Concentration (Cmax) of BAY1143572 after Single Dose Administration in Plasma | Pre-dose up to 24 hours post-dose on Cycle1 Day 1
  Maximum total observed drug concentration of BAY1143572 after single dose administration in plasma was measured.
Maximum Total Observed Drug Concentration of BAY1143572 after Multiple Dose Administration in Plasma (Cmax,md) | Pre-dose up to 24 hours post-dose on Cycle 1 Day 15
  Maximum total observed drug concentration of BAY1143572 after multiple dose administration in plasma was measured.
Area Under the Concentration Versus Time Curve from Zero to 24 hours (AUC[0-24h]) of BAY1143572 in Plasma After Single Dose Administration | Pre-dose up to 24 hours post-dose on Cycle1 Day 1
  Area under the concentration versus time curve from zero to 24 hours of BAY1143572 in plasma after single dose administration was measured.
Area Under the Concentration Versus Time Curve from Zero to 24 hours of BAY1143572 in Plasma after Multiple Dose Administration (AUC[O-24h]md) | Pre-dose up to 24 hours post-dose on Cycle 1 Day 15
  Area under the concentration versus time curve from zero to 24 hours of BAY1143572 in plasma after multiple dose administration was measured.
Area Under the Concentration Versus Time Curve from Zero to Last Data Point Greater than Lower Limit of Quantitation (LLOQ) of BAY1143572 in Plasma (AUC[0-tlast]) after Single Dose Administration | Pre-dose up to 24 hours post-dose on Cycle 1 Day 1
  Area under the concentration versus time curve from zero to last data point greater than lower limit of quantitation of BAY1143572 in plasma after single dose administration was measured.
Time to Reach Maximum Drug Concentration (tmax) of BAY1143572 in Plasma after Single Dose Administration | pre-dose up to 24 hours post-dose on Cycle 1 Day 1
  Time to reach maximum drug concentration of BAY1143572 in plasma after single dose administration was measured.
Time to Reach Maximum Drug Concentration of BAY1143572 in Plasma after Multiple Dose Administration (tmax,md) | Pre-dose up to 24 hours post-dose on Cycle 1 Day 15
  Time to reach maximum drug concentration of BAY1143572 in plasma after multiple dose administration was measured.

SECONDARY OUTCOMES:
Number of Subjects With Leukemia Response | From start of treatment of the first subject until 28 days
  Bone marrow aspirates / biopsies / peripheral whole blood were taken and assessed for leukemia response evaluation. Assessment of response was made based on the revised recommendations of the International Working Group (Cheson 2003 criteria). Criteria proposed by Cheson 2003 for leukemia: complete remission (CR), morphological CR with incomplete blood count recovery (CRi), partial remission (PR), no response / treatment failure, relapse from CR, CRi, or PR.
Number of Subjects with Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | From start of study drug administration up to 30 days after the last dose of study drug administration (approximately 2.5 years)
  An adverse event (AE) was any untoward medical occurrence in subject who received study drug without regard to possibility of causal relationship. AEs that started or worsened after first administration of study medication up to 30 days after end of treatment with study medication were considered to be treatment emergent (TE). A serious adverse event (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly and another medical important serious event as judged by investigator. SAEs that started or worsened after study drug treatment were recorded as TESAEs.
Area Under the Concentration Versus Time Curve from Zero to Infinity (AUC) of BAY1143572 after Single Dose Administration in Plasma | Pre-dose up to 24 hours post-dose on C1D1
  Area under the concentration versus time curve from zero to infinity of BAY1143572 after single dose administration in plasma was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (5):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Germany (2):
  - Universitätsklinikum der Johann Wolfgang Goethe Universität, Frankfurt am Main, Hesse
  - Medizinische Fakultät Carl Gustav Carus, Dresden, Saxony